CLINICAL TRIAL: NCT03785925
Title: A Phase 2, Single-Arm Study of Bempegaldesleukin (NKTR-214) in Combination With Nivolumab in Cisplatin Ineligible, Locally Advanced or Metastatic Urothelial Cancer Patients
Brief Title: A Single-Arm Study of Bempegaldesleukin (NKTR-214) Plus Nivolumab in Cisplatin Ineligible Patients Who Have Locally Advanced or Metastatic Urothelial Cancer
Acronym: PIVOT-10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-214-10; CA045-012 (Other: Bristol-Myers Squibb Protocol ID); 2018-003636-79 (EudraCT Number)
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Urinary Bladder Neoplasm; Neoplasm Metastasis
Keywords: Bladder; Bladder Cancer; CD122; Cisplatin Ineligible; Immuno-oncology; Immunotherapy; Locally Advanced Urothelial Cancer; Metastatic Urothelial Cancer; mUC; Natural Killer Cells; Nivolumab; NKTR-214; Opdivo®; PD-L1; Urothelial Cancer; Urothelial; Metastatic Urothelial Carcinoma; Urothelial Carcinoma; Bempegaldesleukin; BEMPEG; CPI Combination; IL-2
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Metastasis; Carcinoma, Transitional Cell | interventions — bempegaldesleukin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination of bempegaldesleukin (NKTR-214) + nivolumab (Experimental): Participants will receive bempegaldesleukin (NKTR-214) in combination with nivolumab.
  Interventions: Biological: Bempegaldesleukin; Biological: Nivolumab

INTERVENTIONS:
Biological: Bempegaldesleukin — Specified dose on specified days
  Other Names: NKTR-214; BMS-986321
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo®; BMS-936658

SUMMARY:
The main purpose of this study is to evaluate the anti-tumor activity of bempegaldesleukin (NKTR-214) in combination with nivolumab by assessing the objective response rate (ORR) in cisplatin ineligible, locally advanced or metastatic urothelial cancer patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Provide written, informed consent to participate in the study and follow the study procedures
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Measurable disease per RECIST 1.1 criteria
* Histologically or cytologically documented inoperable, locally advanced or metastatic urothelial cell carcinoma (also termed TCC)
* Fresh biopsy or archival tissue
* No prior systemic chemotherapy or investigational agent for inoperable locally advanced or mUC
* Ineligible for cisplatin

Key Exclusion Criteria:

* Patients who have an active, known or suspected autoimmune disease
* Patients must not have received prior IL-2 therapy
* Prior treatment with an anti PD-1, anti PD-L1, or anti cytotoxic T lymphocyte associated protein 4 (anti CTLA-4) antibody, agents that target IL-2 pathway, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Patients with hypertension must be on a stable antihypertensive regimen for the 14 days prior to Cycle 1 Day 1

Additional protocol-defined inclusion/exclusion criteria applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (70):
- United States (8):
  - San Francisco VA Medical Center - NAVREF - PPDS, San Francisco, California
  - Innovative Clinical Research Institute, LLC, Whittier, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Southeastern Regional Medical Center - CTCA - PPDS, Newnan, Georgia
  - Investigator Site - Peoria, Peoria, Illinois
  - Laura And Isaac Perlmutter Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Argentina (7):
  - Centro de Investigación Clínica - Clínica Viedma, Viedma, Río Negro Province
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - CAIPO Centro para la atención integral del paciente oncológico, San Miguel de Tucumán, Tucumán Province
  - Hospital Alemán, Buenos Aires
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires
  - Centro Médico Privado CEMAIC, Córdoba
  - Sanatorio Privado Duarte Quirós, de Clínica Colombo S.A., Córdoba
- Australia (5):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Tasman Health Care, Southport, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Monash Health, Monash Medical Centre, Bentleigh East, Victoria
  - St John of God Murdoch Hospital, Nedlands, Western Australia
- Belgium (3):
  - Algemeen Ziekenhuis Klina, Brasschaat, Antwerpen
  - GasthuisZusters Antwerpen, Wilrijk, Antwerpen
  - AZ Groeninge, Kortrijk
- University Health Network, Toronto, Ontario, Canada
- Helsingin Yliopistollinen Keskussairaala - PPDS, Helsinki, Finland
- France (6):
  - Centre François Baclesse, Caen, Calvados
  - Hôpital Privé TOULON/HYERES Sainte Marguerite, Hyères
  - Centre Jean Bernard Clinique Victor Hugo, Le Mans
  - Hôpital Européen Georges Pompidou, Paris
  - Edog Ico - Ppds, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - Kliniken Nordoberpfalz AG, Weiden, Bavaria
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
- Greece (4):
  - Alexandra Hospital, Athens, Attica
  - Medical Center of Athens, Marousi, Attica
  - University General Hospital of Larissa, Larissa
  - Euromedica - PPDS, Thessaloniki
- Israel (5):
  - Shamir Medical Center Assaf Harofeh, Ẕerifin, Central District
  - Rambam Medical Center - PPDS, Haifa
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center - PPDS, Ramat Gan
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (3):
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST - PPDS, Meldola, Emilia-Romagna
  - Centro Di Riferimento Oncologico, Aviano, Pordenone
  - Istituto Nazionale Dei Tumori, Milan
- Mexico (2):
  - Health Pharma Professional Research S.A de C.V., Mexico City, Mexico City
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli
- Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- Centro Hospitalar E Universitário de Coimbra EPE, Coimbra, Portugal
- Russia (5):
  - Regional Clinical Oncology Hospital, Yaroslavl, Yaroslavl Oblast
  - Federal State Institution Medical Radiology Research Center, Obninsk
  - Clinical Oncology Dispensary, Omsk
  - PMI Euromedservice, Pushkin
  - Railway Clinical Hospital JSC RZhD, Saint Petersburg
- Spain (8):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de La Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Ramon y Cajal, Pozuelo de Alarcón, Madrid
  - Hospital del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- Turkey (Türkiye) (3):
  - Ankara University Medical Faculty - PPDS, Ankara
  - Izmir Medicalpark Hospital, Izmir
  - Inonu University Faculty of Medicine Turgut Ozal Medical Center, Malatya
- United Kingdom (3):
  - Royal Marsden Hospital - Surrey, Sutton, Surrey
  - Leicester Royal Infirmary, Leicester
  - Barts Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 192 patients were enrolled. Two patients withdrew consent before treatment. Two patients received Gemcitabine + Carboplatin under protocol amendment 2.0. The noncomparative, reference chemotherapy arm of gemcitabine + carboplatin was subsequently eliminated in protocol amendment 3.0. These four patients were excluded from the analysis.
Groups:
- Combination of Bempegaldesleukin (NKTR-214) + Nivolumab: Participants received bempegaldesleukin (NKTR-214) at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
  The Treated Population included 188 patients; from these, 123 had tumors with low PD-L1 expression, 59 had tumors with high PD-L1 expression, and 6 had unknown PD-L1 expression.
Period: Overall Study
Arm/Group | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab
Started | 188
Completed | 172
Not Completed | 16
Not completed — Withdrawal by Subject | 15
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of 188 patients.
Groups:
- Combination of Bempegaldesleukin (NKTR-214) + Nivolumab: Participants received bempegaldesleukin (NKTR-214) at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
Arm/Group | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab
Number analyzed (Participants) | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8.21)
Age, Customized [Count of Participants; unit: Participants]
  Age < 65 | 37
  Age 65-84 | 141
  Age 85 and Over | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 155
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 171
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  Argentina | 14
  United States | 36
  United Kingdom | 6
  Portugal | 2
  Russia | 21
  Spain | 27
  Greece | 10
  Canada | 3
  Netherlands | 6
  Turkey | 8
  Belgium | 5
  Finland | 2
  Italy | 8
  Mexico | 1
  Israel | 11
  Australia | 14
  France | 9
  Germany | 5
ECOG Performance Status [Count of Participants; unit: Participants] — Measure Description: Eastern Cooperative Oncology Group (ECOG) performance status:
  ECOG Performance Status of 0 = Able to carry out all normal activities without restriction ECOG Performance Status of 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature
  Participants
    ECOG PS 0 | 64
    ECOG PS 1 | 73
    ECOG PS 2 | 51

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Per Blinded Independent Central Review (BICR) in Patients Whose Tumors Have Low Programmed Cell Death Ligand (PD-L1) Expression
Description: To evaluate the anti-tumor activity of NKTR-214 in combination with nivolumab by assessing the ORR by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) per blinded independent central review (BICR) in patients whose tumors have low programmed cell death ligand 1 (PD-L1) expression. ORR was defined as the percentage of patients with confirmed objective response of Complete Response (CR) or Partial Response (PR) on or before the first progressive disease and any subsequent anticancer therapy.
  CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumor assessments were performed at baseline and every 9 weeks from Cycle 1 Day 1 for the first 12 months, and then every 12 weeks as indicated in the Schedule of Events, up to approximately 27 months
Population: The primary endpoint of ORR per RECIST 1.1 by BICR was evaluated in the Treated PD-L1 Low Population (123 patients).
  The Treated Population included 188 patients who were enrolled and received at least one full (or partial dose) of NKTR-214 or nivolumab.
  PD-L1 Low: Patients in the Treated Population whose tumors had low PD-L1 expression (defined as Combined Positive Score [CPS] < 10). From the 188 patients, 123 had tumors with low PD-L1 expression.
Measure: Count of Participants; unit: Participants
Groups:
- PD-L1 Low: ORR per RECIST 1.1 by BICR in PD-L1 Low Patients
Arm/Group | PD-L1 Low
Number analyzed (Participants) | 123
Participants | 22

2. Secondary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Per Blinded Independent Central Review (BICR) in All Treated Patients
Description: To evaluate the anti-tumor activity of NKTR-214 in combination with nivolumab by assessing the ORR by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) per blinded independent central review (BICR) in all treated patients. ORR was defined as the percentage of patients with confirmed objective response of Complete Response (CR) or Partial Response (PR) on or before the first progressive disease and any subsequent anticancer therapy.
  CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 1
Population: The secondary endpoint of ORR per RECIST 1.1 by BICR was evaluated in the Treated Population (188 patients).
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab
Number analyzed (Participants) | 188
Participants | 37

3. Secondary Outcome: Duration of Response (DOR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Per Blinded Independent Central Review (BICR) in in All Treated Patients and Patients Whose Tumors Have Low Programmed Cell Death Ligand (PD-L1) Expression
Description: To evaluate the effect of NKTR 214 in combination with nivolumab by assessing DOR by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) per blinded independent central review (BICR) in all treated patients and patients whose tumors have low PD-L1 expression.
  DOR is defined for patients who have a confirmed Complete Response (CR) or Partial Response (PR) as the date from first documented CR or PR per RECIST 1.1 to the date of documentation of disease progression as assessed by BICR or death due to any cause, whichever is earlier. Patients who do not have disease progression or die will be censored on the date of their last evaluable tumor assessment.
Time Frame: as for outcome 1
Population: All Treated Population who had a confirmed Complete Response (CR) or Partial Response (PR) per RECIST 1.1.
  Treated PD-L1 Low: Patients in the Treated Population whose tumors had low PD-L1 expression (defined as Combined Positive Score [CPS] < 10).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (All Treated Population): Participants received bempegaldesleukin (NKTR-214) at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
- Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (PD-L1 Low Population): Arm Group Description: Participants received bempegaldesleukin (NKTR-214) at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
Arm/Group | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (All Treated Population) | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (PD-L1 Low Population)
Number analyzed (Participants) | 37 | 22
Months | 13.4 [8.2 to NA] — NA = 95% CI upper limit could not be estimated due to an insufficient number of participants | 13.4 [6.2 to NA] — NA = 95% CI upper limit could not be estimated due to an insufficient number of participants

4. Secondary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Investigator in All Treated Patients and Patients Whose Tumors Have Low Programmed Cell Death Ligand (PD-L1) Expression
Description: To evaluate the anti-tumor activity of NKTR-214 in combination with nivolumab by assessing the ORR by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) by Investigator Assessment in All Treated Patients and Patients Whose Tumors Have Low Programmed Cell Death Ligand (PD-L1) Expression.
  ORR was defined as the percentage of patients with confirmed objective response of Complete Response (CR) or Partial Response (PR) on or before the first progressive disease and any subsequent anticancer therapy.
Time Frame: as for outcome 1
Population: The All Treated Population included 188 patients who were enrolled and received at least one full (or partial dose) of NKTR-214 or nivolumab.
  Treated PD-L1 Low: Patients in the Treated Population whose tumors had low PD-L1 expression (defined as Combined Positive Score [CPS] < 10). From the 188 patients, 123 had tumors with low PD-L1 expression.
Measure: Count of Participants; unit: Participants
Groups:
- Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (All Treated Population): Participants received bempegaldesleukin (NKTR-214) at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
  The Treated Population included 188 patients.
- Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (PD-L1 Low Population): Arm Group Description: Participants received bempegaldesleukin (NKTR-214) at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
  The PD-L1 Low Population included 123 patients.
Arm/Group | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (All Treated Population) | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (PD-L1 Low Population)
Number analyzed (Participants) | 188 | 123
Participants | 36 | 20

5. Secondary Outcome: Duration of Response (DOR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Investigator in All Treated Patients and Patients Whose Tumors Have Low Programmed Cell Death Ligand (PD-L1) Expression
Description: To evaluate the effect of NKTR 214 in combination with nivolumab by assessing DOR by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) by Investigator Assessment in all treated patients and patients whose tumors have low PD-L1 expression.
  DOR is defined for patients who have a confirmed Complete Response (CR) or Partial Response (PR) as the date from first documented CR or PR per RECIST 1.1 to the date of documentation of disease progression as assessed by BICR or death due to any cause, whichever is earlier. Patients who do not have disease progression or die will be censored on the date of their last evaluable tumor assessment.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (All Treated Population) | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (PD-L1 Low Population)
Number analyzed (Participants) | 36 | 20
Months | 15.9 [10.7 to NA] — NA = 95% CI upper limit could not be estimated due to an insufficient number of participants | 14.3 [8.2 to NA] — NA = 95% CI upper limit could not be estimated due to an insufficient number of participants

ADVERSE EVENTS:
Time Frame: AEs were reported from the time of first study drug(s) administration until 100 days after the last dose of all study drug(s), up to a maximum of approximately 27 months.
Arm/Group | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab
All-Cause Mortality (participants affected / at risk) | 127/188
Serious Adverse Events (participants affected / at risk) | 98/188
Other Adverse Events (participants affected / at risk) | 185/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (N=188)
Urinary tract infection (Infections and infestations) | 12
Acute kidney injury (Renal and urinary disorders) | 9
Haematuria (Renal and urinary disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Pyrexia (General disorders) | 5
Pneumonia (Infections and infestations) | 4
Urosepsis (Infections and infestations) | 4
Corona virus infection (Infections and infestations) | 3
Fatigue (General disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Urinary tract infection enterococcal (Infections and infestations) | 2
Hydronephrosis (Renal and urinary disorders) | 2
Nephritis (Renal and urinary disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
General physical health deterioration (General disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Myocarditis (Cardiac disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Peripheral ischaemia (Vascular disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 2
Bacterial sepsis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Pyelonephritis chronic (Infections and infestations) | 1
Renal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Spinal cord infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Vascular device infection (Infections and infestations) | 1
Bladder neck obstruction (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Kidney congestion (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract discomfort (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Sudden death (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebral microembolism (Nervous system disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Scrotal pain (Reproductive system and breast disorders) | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Hypophysitis (Endocrine disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Device occlusion (Product Issues) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (N=188)
Pyrexia (General disorders) | 82
Fatigue (General disorders) | 58
Decreased appetite (Metabolism and nutrition disorders) | 58
Anaemia (Blood and lymphatic system disorders) | 57
Diarrhoea (Gastrointestinal disorders) | 56
Nausea (Gastrointestinal disorders) | 54
Constipation (Gastrointestinal disorders) | 44
Pruritus (Skin and subcutaneous tissue disorders) | 43
Pruritus generalised (Skin and subcutaneous tissue disorders) | 40
Urinary tract infection (Infections and infestations) | 39
Asthenia (General disorders) | 36
Vomiting (Gastrointestinal disorders) | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 35
Oedema peripheral (General disorders) | 32
Haematuria (Renal and urinary disorders) | 31
Hypothyroidism (Endocrine disorders) | 28
Chills (General disorders) | 27
Eosinophilia (Blood and lymphatic system disorders) | 26
Blood creatinine increased (Investigations) | 25
Influenza like illness (General disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 23
Dizziness (Nervous system disorders) | 22
Hypotension (Vascular disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Rash (Skin and subcutaneous tissue disorders) | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Headache (Nervous system disorders) | 19
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17
Hyperthyroidism (Endocrine disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 15
Rash generalised (Skin and subcutaneous tissue disorders) | 15
Gamma-glutamyltransferase increased (Investigations) | 15
Insomnia (Psychiatric disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Weight decreased (Investigations) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13
Hyponatraemia (Metabolism and nutrition disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Blood alkaline phosphatase increased (Investigations) | 12
Infusion related reaction (Injury, poisoning and procedural complications) | 12
Dry mouth (Gastrointestinal disorders) | 11
Amylase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 11
Hypertension (Vascular disorders) | 11
Face oedema (General disorders) | 10
Alanine aminotransferase increased (Investigations) | 10
Fall (Injury, poisoning and procedural complications) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.

DOCUMENTS (2):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT03785925/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT03785925/SAP_001.pdf